CLINICAL TRIAL: NCT04003454
Title: The Determining Effective Testing in Emergency Departments and Care Coordination on Treatment Outcomes (DETECT) for HCV Trial
Brief Title: The DETECT HCV Screening Trial
Acronym: DETECT HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Johns Hopkins University (Other); University of Mississippi Medical Center (Other); Boston University (Other); Boston Medical Center (Other); University of Cincinnati (Other); Alameda County Medical Center (Other)
Responsible Party: Principal Investigator, Jason Haukoos, Professor & Director of Research, Department of Emergency Medicine, Denver Health, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01DA042982 (NIH)
Record Dates: First submitted 2019-04-05; First posted 2019-07-01 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Screening; Emergency Department; Risk
MeSH Terms: conditions — Hepatitis C; Emergencies

STUDY DESIGN:
Intervention Model Description: Patients presenting to the emergency department will be randomized to targeted HCV screening or nontargeted HCV screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nontargeted Screening (Other): The nontargeted HCV screening arm will consist of implementing non-risk-based rapid opt-out HCV screening.
  Interventions: Other: HCV Screening
- Targeted Screening (Other): The targeted HCV screening arm will consist of implementation of risk-based rapid opt-out HCV screening using current recommendations for HCV screening by the CDC, USPSTF, and AASLD-IDSA. Targeted HCV screening will consist of offering HCV testing to those identified with the following specific risk characteristics, adapted from the above recommendations: born between 1945 - 1965 ("birth cohort"); injection drug use (IDU); intranasal drug use;tattoo or piercing in an unregulated setting; or blood transfusion or organ recipient before 1992.
  Interventions: Other: HCV Screening

INTERVENTIONS:
Other: HCV Screening — The investigators will perform a prospective pragmatic randomized effectiveness trial that will allow the investigators to directly compare 2 HCV screening methods while minimizing threats to internal validity. Patients will be screened for HCV infection using 1 of 2 interventions using a balanced patient-level random allocation scheme built into existing EHRs for each ED.

SUMMARY:
The investigators propose to compare the effectiveness of nontargeted rapid opt-out hepatitis C (HCV) screening versus targeted rapid opt-out HCV screening using recommended risk characteristics in multiple urban emergency departments (EDs) across the United States (Aim 1 - "Screening Trial").

DETAILED DESCRIPTION:
The investigators will perform a prospective pragmatic randomized effectiveness trial that will allow the investigators to directly compare 2 HCV screening methods while minimizing threats to internal validity. Patients will be screened for HCV infection using 1 of 2 interventions using a balanced patient-level random allocation scheme built into existing electronic health records (EHRs) for each ED. Patients will therefore be offered HCV testing based on the result of the screening arm to which they are assigned, and in the case of the targeted arm, the results of the risk assessment evaluation performed by the intake nurse. All randomization will be completely integrated into electronic medical screening systems and workflow at each site. Integration of randomization into the electronic systems will allow for real-time concealed random allocation. Nurses who perform screening and all other ED staff (e.g. physicians, technicians) will understand the conceptual goals of the project but will be blinded to study hypotheses, and patients will be completely blinded to the purpose of the study.

This study will be performed at multiple sites, including the EDs at Denver Health Medical Center (DHMC) (Denver, Colorado), Johns Hopkins Hospital (JHH) (Baltimore, Maryland), and the University of Mississippi Medical Center (UMMC) (Jackson, Mississippi).

ELIGIBILITY:
Inclusion Criteria:

* Present to EDs during study enrollment period
* Clinically stable per screening nurse or physician assessment
* Able to provide consent for medical care

Exclusion Criteria:

* Younger than 18 years of age
* Are unable to consent for care (i.e., altered mentation, critical illness, or injury)
* Have already participated in the trial
* Self-Identify as already living with HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147533 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Newly diagnosed active HCV | 1 day from ED visit
  Confirmed cases of newly diagnosed active HCV, defined as patients who test positive for HCV antibody and measurable HCV RNA, and without a prior HCV diagnosis, stratified by study arm

SECONDARY OUTCOMES:
HCV test acceptance | 1 day from ED visit
  Defined by the proportion of patients who agree to HCV testing, as measured by the proportion of those who consent among patients offered HCV testing, stratified by study arm
HCV test completion | 1 day from ED visit
  Defined by the proportion of patients who complete HCV testing, as measured by the proportion of rapid HCV tests completed among patients who accepted testing, stratified by study arm

OTHER OUTCOMES:
HCV genotype among those identified with active HCV | 12 months following HCV diagnosis
  Measured by HCV genotyping among those identified with active HCV
Fibrosis staging | 12 months following HCV diagnosis
  Measured by standard of care fibrosis staging approaches (e.g. biopsy, ultrasound, FibroTest, etc.) among those identified with active HCV
Completion of an evaluation by an HCV treatment expert | 12 months following HCV diagnosis
  Measured by indication of a completed visit with an HCV treatment expert among those identified with active HCV
Initiation of treatment with Direct-Acting Antivirals (DAAs) | 12 months following HCV diagnosis
  Measured by indication of initiation of treatment with DAAs among those identified with active HCV
Completion of treatment with Direct-Acting Antivirals (DAAs) | 12 months following HCV diagnosis
  Measured by indication of completion of treatment with DAAs among those identified with active HCV
Sustained virologic response at 12 weeks after treatment completion (SVR12) | 12 months following HCV diagnosis
  Measured by undetectable HCV RNA 12 weeks after completion of DAAs among those identified with active HCV

CONTACTS AND LOCATIONS:
Overall Officials: Jason Haukoos, MD, MSc, Principal Investigator — Denver Health; Sarah Rowan, MD, Principal Investigator — Denver Health
Locations (3):
- United States (3):
  - Denver Health Medical Center, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haukoos J, Rothman RE, Galbraith JW, Hopkins E, Hsieh YH, Lyle C, Gravitz S, Kamis KF, White DAE, Lyons MS, Gardner EM, Al-Tayyib AA, Sabel AL, Linas BP, Morgan JR, Wyles DL, Rowan SE; DETECT Hep C Screening Trial Investigators. Hepatitis C Screening in Emergency Departments: The DETECT Hep C Randomized Clinical Trial. JAMA. 2025 Aug 12;334(6):497-507. doi: 10.1001/jama.2025.10563. PMID 40632510
- [Derived] Haukoos JS, Rowan SE, Galbraith JW, Rothman RE, Hsieh YH, Hopkins E, Houk RA, Toerper MF, Kamis KF, Morgan JR, Linas BP, Al-Tayyib AA, Gardner EM, Lyons MS, Sabel AL, White DAE, Wyles DL; DETECT Hep C Trials Investigators. The Determining Effective Testing in Emergency Departments and Care Coordination on Treatment Outcomes (DETECT) for Hepatitis C (Hep C) Screening Trial: rationale and design of a multi-center pragmatic randomized clinical trial of hepatitis C screening in emergency departments. Trials. 2022 Apr 25;23(1):354. doi: 10.1186/s13063-022-06265-1. PMID 35468807